CLINICAL TRIAL: NCT06449001
Title: A Phase 3 Open-Label Study of Danicopan as Add-on Treatment to Ravulizumab or Eculizumab in Pediatric Participants With Paroxysmal Nocturnal Hemoglobinuria Who Have Clinically Significant Extravascular Hemolysis
Brief Title: Study of Danicopan as Add-on Treatment to Ravulizumab or Eculizumab in Pediatric Participants With PNH Who Have Clinically Significant Extravascular Hemolysis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7332C00006; ALXN2040-PNH-302 (Other: Alexion)
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria; PNH; Extravascular Hemolysis
Keywords: Paroxysmal Nocturnal Hemoglobinuria; PNH; Extravascular Hemolysis; Ravulizumab; Eculizumab; Danicopan
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Hemolysis | interventions — danicopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Danicopan (Experimental): Participants will receive a 12-week weight-based open-label treatment period and up to 1 year open-label long term extension period.
  Interventions: Drug: Danicopan

INTERVENTIONS:
Drug: Danicopan — Participants will receive danicopan on a weight-based dosing regimen.

SUMMARY:
The primary objective of this study is to evaluate efficacy of danicopan as add-on treatment to ravulizumab or eculizumab as assessed by hemoglobin (Hgb) change from Baseline at Week 12 in pediatric participants with paroxysmal nocturnal hemoglobinuria (PNH) and clinically significant extravascular hemolysis (CS-EVH).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PNH.
* CS-EVH defined by: Anemia: Hgb ≤ 11.0 g/dL, and absolute reticulocyte count ≥ 100 × 109/L
* Treated with ravulizumab or eculizumab for at least 12 weeks immediately preceding Day 1, the dose received should be stable during this period, and there should be no anticipated changes in dosage or interval during the first 12 weeks of this study.
* all participants must be vaccinated against meningococcal infection from serogroups A, C, W, and Y and serogroup B within 3 years prior to, or at least 14 days prior to Day 1
* vaccinated against Haemophilus influenzae type b (Hib) and Streptococcus pneumoniae

Exclusion Criteria:

* Platelet count < 30000/μL or there is a need for platelet transfusions.
* ANC < 500/μL.
* Clinically significant laboratory abnormalities related to liver function, including:

  * ALT > 2 × ULN or ALT > 3 × ULN for participants with documented liver iron overload defined by serum ferritin values ≥ 500 ng/mL.
  * Direct bilirubin > 2 × ULN, unless, in the Investigator's opinion, is due to hemolysis or Gilbert's syndrome based on medical history.
* Current evidence of biliary cholestasis.
* Known aplastic anemia or other bone marrow failure that requires HSCT or other therapies, including anti-thymocyte globulin and immunosuppressants unless the dosage of immunosuppressant has been stable for at least 12 weeks before Day 1 and is expected to remain stable through Week 12.
* History of a major organ transplant (eg, heart, lung, kidney, liver) or HSCT.
* Known or suspected complement deficiency.
* Active bacterial or viral infection, a body temperature > 38°C on 2 consecutive daily measures, evidence of other infection, or history of any febrile illness within 14 days prior to first study intervention administration.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2027-05-28 (Estimated); Study Completion 2028-03-10 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Hemoglobin (Hgb) Concentration at Week 12 | Baseline, Week 12

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Danicopan | Day 1 up to Week 12
Number of Participants With Transfusion Avoidance Through Weeks 12 and 24 | Weeks 12 and 24
Change From Baseline in Absolute Reticulocyte Count at Weeks 12 and 24 | Baseline, Weeks 12 and 24
Change From Baseline in Pediatric Quality of Life Inventory (PedsQL) Generic Core Scales Score at Weeks 12 and 24 | Baseline, Weeks 12 and 24
Change from Baseline in Pediatric Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score at Weeks 12 and 24 | Baseline, Weeks 12 and 24
Acceptability and Palatability Questionnaire Score | Week 2
Change from Baseline in Hgb Concentration at Week 24 | Baseline, Week 24
Change from Baseline in Serum Alternative Pathway (AP) Activity | Baseline up to Week 64
Change from Baseline in Plasma Bb Concentrations | Baseline up to Week 64

CONTACTS AND LOCATIONS:
Locations (4):
- Research Site, Saskatoon, Saskatchewan, Canada
- Research Site, Paris, France
- United Kingdom (2):
  - Research Site, Leeds
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR